CLINICAL TRIAL: NCT04463810
Title: The Evaluations of Cardiovascular Changes in Long-term Treated HIV-infected Chinese Individuals
Brief Title: The Evaluations of Cardiovascular Changes in Long-term Treated HIV-infected Individuals
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LI Taisheng, Chief, Department of Infectious Diseases, Peking Union Medical College Hospital
Other Study IDs: CACT1808
Record Dates: First submitted 2018-07-15; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: HIV/AIDS; Cardiovascular Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study aims to evaluate the cardiovascular changes in long-term virologically controlled HIV patients. All the participants have been treated and have been undetected for at least five years. Vascular ultrasound and echo will be carried out at 0, 24, 48 and 96 weeks of follow-up.

DETAILED DESCRIPTION:
Previous studies have indicated that chronic HIV infection has resulted the diastolic cardiac dysfunction. In this study, 500 long-term virologically controlled HIV-infected individuals will be followed for two years, and evaluated at 0, 24, 48 and 96 weeks of follow-up. At each visiting point, ultrasound evaluation of carotid and vertebral arteries and the heart function will be carried out and compared.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Willingness and availability to engage in study activities for the duration of the study
* Age between 18-65
* Documented HIV-1 infection (confirmed by Western blot)
* regular ART treated for over 240 weeks
* HIV-RNA < 200 cp/ml

Exclusion Criteria:

* Pregnancy or breastfeeding or anticipated pregnancy in two years
* History of AIDS-defining illness
* Virological failure during the ART ( Definition of virolgocial failure: plasma HIV-RNA > 200 cp/ml upon continuous HARRT)
* Hemoglobin < 9g/dl；or peripheral white blood cell counts < 2000/μl；or neutrophil counts < 1000 /μl；or platelet count < 75,000/μl；
* Liver disease (transaminase and alkaline phosphatase levels more than three times the upper limit of the normal range (ULN), bilirubin level more than 2.5 times the ULN)
* Chronic kidney disease (serum creatinine level more than 1.5 times the ULN)
* Patients with a history of injection drug usage
* Patients with a history of mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: long-term treated HIV-infected patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with abnormal brachial-ankle arteries measured by ultrasound at 48 weeks | 48 weeks
  The ankle-brachial index (ABI) and pulse wave velocity (PWV) including right and left brachial-ankle are aceessed through ultrasound. The measured value will be documented and evaluated for abnormality.
Number of Participants with abnormal brachial-ankle arteries measured by ultrasound at 96 weeks | 96 weeks
  The ankle-brachial index (ABI) and pulse wave velocity (PWV) including right and left brachial-ankle are aceessed through ultrasound. The measured value will be documented and evaluated for abnormality.
Number of Participants with abnormal echocardiogram results at 48 weeks | 48 weeks
  Echocardiogram indicators include left ventricular end-diastolic diameter, left ventricular end-systolic diameter, left ventricular fractional shortening (LVFS), ejection fraction (EF), E/A ratio, E-wave deceleration time (EDT), isovolumetric relaxation time (IVRT), tricuspid regurgitation velocity (TRV), Pulmonary artery systolic pressure, Interventricular septal (IVS ) thickness, left ventricular posterior wall thickness, the present of valve abnormalities/ myocardial ischemia/ pericardial effusion. The measured value will be documented and evaluated for abnormality.
Number of Participants with abnormal echocardiogram results at 96 weeks | 96 weeks
  Echocardiogram indicators include left ventricular end-diastolic diameter, left ventricular end-systolic diameter, left ventricular fractional shortening (LVFS), ejection fraction (EF), E/A ratio, E-wave deceleration time (EDT), isovolumetric relaxation time (IVRT), tricuspid regurgitation velocity (TRV), Pulmonary artery systolic pressure, Interventricular septal (IVS ) thickness, left ventricular posterior wall thickness, the present of valve abnormalities/ myocardial ischemia/ pericardial effusion. The measured value will be documented and evaluated for abnormality.

SECONDARY OUTCOMES:
Changes from baseline T cellular activation markers | 0,24,48 and 96weeks
  Changes from baseline T cellular activation markers (CD8CD38+ T percentage and CD8DR+ T percentage).
Changes from baseline serum inflammatory markers | 0,24,48 and 96weeks
  Changes from baseline serum inflammatory markers (sCD14, D-dimer, IL-6, IP-10)

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided